CLINICAL TRIAL: NCT00115843
Title: Atrial Fibrillation Rate Control Therapy Guided By Continuous Ambulatory Monitoring
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Cardionet (Industry)
Responsible Party: Principal Investigator, Peter Zimetbaum, Richard A. and Susan F. Smith Professor of Medicine in the Field of Cardiovascular Medicine, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2004P000346
Record Dates: First submitted 2005-06-26; First posted 2005-06-27 (Estimated); Last update posted 2017-04-05 (Actual); Status verified 2017-04

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; Arrhythmia; Tachycardia
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac; Tachycardia

INTERVENTIONS:
Device: Mobile Cardiac Outpatient Telemetry

SUMMARY:
The purpose of this study is to demonstrate that the use of a continuous ambulatory monitoring device will reduce both the time to effective rate control and the health care expenditures associated with standard methods of rate control monitoring in patients presenting with atrial fibrillation with a rapid heart rate.

DETAILED DESCRIPTION:
This is an open, randomized controlled trial to compare a standard rate-control strategy with one using the Cardionet device to guide therapy for the management of atrial fibrillation. Patients presenting to an outpatient clinic or to the Emergency Department with atrial fibrillation with a ventricular rate greater than 100 bpm at rest will be enrolled.

Treatment:

Patients will be prescribed either a beta blocker or a calcium channel blocker, or have their baseline dose increased if already taking one of these agents at the discretion of the treating physician. This is consistent with standard outpatient treatment guidelines for rate control in atrial fibrillation.

Randomization:

At the time of enrollment, patients will be randomized to a standard rate control protocol or a rate-control protocol guided by the Cardionet device.

Standard Care (Comparison Group):

Patients randomized to standard care will have a home patient educator install the Cardionet device within 24 hours after enrollment. The Cardionet device will be used to adjudicate the primary endpoint of adequate rate control in the standard care group. The patient's treating physician will be blinded to the reports from the Cardionet device. These patients will have another office visit with the initial referring physician or a staff cardiologist within the first week after enrollment and weekly thereafter. At this time, adequacy of rate control will be assessed by a standard 12-lead electrocardiogram and patient history. Medication will be adjusted per protocol. The patient will be seen on a weekly basis until adequate rate control is thought to have been achieved.

Rate Control using Cardionet (Study Group):

Patients randomized to use of the Cardionet device will have a home patient educator install the device within 24 hours after enrollment. Electrocardiographic summaries will be reviewed by a research physician three times a week and treatment decisions will be made based on a summary of 24-hour rate control. The physician will contact the patient by telephone and make medication adjustments per protocol. Three-times-weekly transmissions and medication adjustments will continue until adequate rate control is achieved over a period of 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Atrial fibrillation with resting ventricular rate > 100 with rate control strategy indicated
* Atrial fibrillation is likely to be recurrent or persistent in the clinical judgment of the physician
* Patient able to be managed out of the hospital
* Ability to sign informed consent
* Ability to wear electrodes for the Cardionet device
* Patient willing to have home patient educator install Cardionet monitor in their home

Exclusion Criteria:

* Inability to follow up with prescribed schedule of monitoring
* Concomitant use of antiarrhythmic drug
* Indication for hospitalization

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-04; Primary Completion 2006-09; Study Completion 2006-09

PRIMARY OUTCOMES:
Time to adequate heart rate (HR) control, defined as resting heart rate ≤ 80 bpm and average heart rate over 24 hours < 100 and no recorded HR > 110% of maximum age-adjusted predicted HR.

SECONDARY OUTCOMES:
Total health care costs associated with conventional and Cardionet based monitoring strategy.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Zimetbaum, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States